CLINICAL TRIAL: NCT06704061
Title: Online Yoga vs Acceptance and Commitment Therapy for Treating Chronic Musculoskeletal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Peter Bayley, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAYNEW0004
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: chronic pain; veteran; musculoskeletal pain; yoga
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain | interventions — Yoga; Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Yoga (Experimental): Postures, meditation, breathing exercises
  Interventions: Behavioral: Yoga
- Acceptance and Commitment Therapy (Active Comparator): Behavioral medicine
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)

INTERVENTIONS:
Behavioral: Yoga — A 12-week online yoga course designed to treat pain.
  Arms: Online Yoga
Behavioral: Acceptance and Commitment Therapy (ACT) — A 12-week behavioral therapy course designed to treat pain.
  Arms: Acceptance and Commitment Therapy

SUMMARY:
This study will compare online yoga with Acceptance and Commitment Therapy (ACT), an established treatment for chronic pain. We will compare the efficacy of the two treatments for reducing chronic musculoskeletal pain in veterans.

DETAILED DESCRIPTION:
This study will test if online yoga is not inferior than ACT for treating chronic pain in veterans. Participants will be randomly assigned to receive either online yoga instruction or ACT, once a week for 12 weeks in an online group class. They will complete self-report questionnaires about their experience of chronic pain. There will be a 6-month follow up period, during which the research team will check in with the participant to record any adverse events and maintain study contact.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the United States Armed Forces ≥ 18 years old
* Chronic pain > 6 months related to at least one musculoskeletal pain-related diagnosis indicated by an ICD-9 or -10 code
* Minimum pain intensity at screening ≥4 on a 0-10 using the Defense and Veterans Pain Rating Scale (DVPRS)
* Not begun new pain treatments or medications in the past month
* Stable medication regimen for at least 4 weeks prior to entry to the study
* English literacy
* Internet connection at home

Exclusion Criteria:

* Participation in another clinical trial, unless given prior authorization from both our research team and that of the other study
* Back surgery within the last 12 months
* Back pain potentially attributed to a specific known condition
* Baseline pain <4 or ≥9 on a 0-10 Numeric Rating Scale
* Unstable, serious coexisting medical illness, mental illness or psychiatric conditions
* Attended or practiced yoga ≥ 1 x in the past 12 months
* Current suicidal intent or plan
* Has received ACT in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain Interference (Brief Pain Inventory-Short Form) | Baseline, End-of-treatment at 12 weeks, and 6 months after treatment
  The degree to which pain impacts mood, walking and other daily activities, as measured by the Pain Interference Scale of the Brief Pain Inventory - Short Form (BPI-SF). The BPI-SF assesses intensity and impact of pain on functioning on a 0-10 rating scale, with higher scores indicating greater degree of interference.

SECONDARY OUTCOMES:
Depression (BDI-II) | Baseline, End-of-treatment at 12 weeks, and 6 months after treatment
  Symptoms of depression as measured by the Beck Depression Inventory (BDI-II). The BDI-II is comprised of 21 self-report questions, scored on a 0-3 scale, with higher scores indicating more depressive symptoms.
Sleep (Pittsburgh Sleep Quality Index) | Baseline, End-of-treatment at 12 weeks, and 6 months after treatment
  Sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month interval.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bayley, PhD, Principal Investigator — Palo Alto Veterans Institute for Research
Locations (1):
- Palo Alto VA Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All demographic, clinical observations, and clinical self-reports
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available at the end of the funding period. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: Data and source materials will be posted on DRYAD, an open-source tool for data publication and digital preservation. DRYAD provides searchable study-level metadata for dataset discovery. Data will be indexed by Google Dataset Search and other tools to enhance discoverability and will be discoverable online through standard web search of the study-level metadata as well as the persistent pointer from the DOI to the dataset.